CLINICAL TRIAL: NCT01354041
Title: A Pilot Intervention to Address Fear of Recurrence in Breast Cancer Survivors
Brief Title: Fear of Recurrence Pilot Intervention for Women With Breast Cancer
Acronym: WiLLoW
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-01831
Record Dates: First submitted 2011-02-24; First posted 2011-05-16 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Cancer Recurrence
Keywords: fear and health worries about cancer recurrence
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment-as-usual (No Intervention): Participants in the Treatment as usual (TAU) arm will not receive any specific Fear of Cancer Recurrence (FCR) intervention during the study period. However, they will be offered an optional full-day workshop at the end of the study.
- Acceptance and Commitment Therapy (Experimental): Participants in the intervention arm will receive seven sessions of a mindfulness and values-based living intervention, led by a trained licensed facilitator, conducted in groups of 10-12 participants and include components specifically designed to reduce FCR. The intervention arm will include six weekly 90 minute group sessions and one followup 90 minute group session "booster session" held three weeks later. The group sessions will be interactive and experiential and include homework practice for generalizing skills.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Seven weekly sessions of Acceptance and Commitment Therapy (ACT) intervention
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy

SUMMARY:
The primary objective of this pilot study is to examine the feasibility and acceptability of a randomized, controlled study of a mindfulness and values-based living intervention targeted at reducing fear of recurrence in breast cancer survivors compared to treatment as usual control. Furthermore, the secondary objective of this randomized, controlled pilot study is to determine preliminary efficacy and effect size of the mindfulness and values-based living intervention compared to the treatment as usual control condition in reducing fear of recurrence in breast cancer survivors.

DETAILED DESCRIPTION:
Fear of cancer recurrence (FCR) is pervasive, distressing and undermines quality of life in cancer survivors. For subgroups of survivors, FCR is implicated in both treatment non-adherence and medical over-utilization. Although some degree of FCR is nearly universal among cancer patients, effective psychological interventions have been understudied. Educational and cognitive approaches that have relied on reassurance may feed into the anxiety by encouraging experiential avoidance, according to behavioral theories of anxiety. Mindfulness and values based living approaches teach techniques for reducing experiential avoidance allowing patients to break this cycle and focus on functional, satisfying lives. Interventions based on these techniques offer promise for addressing FCR in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage breast cancer within the past 18 months;
* Completed active treatment within the past year
* At least mild anxiety, and/or at least moderate fear of recurrence as measured by screening questionnaires.
* Ability to give written informed consent and willingness to comply with the requirements of the protocol

Exclusion Criteria:

* Presence of clinically significant cognitive impairment, or comorbid psychiatric or physical illness, only if, in the PI's or Co-Is' opinions, such illness would interfere with the ability to participate in and complete the intervention;
* Inability to speak and comprehend English sufficiently to complete the intervention.
* We will use a screening questionnaire (administered over the phone by the Research Associate) to determine that women do not have a comorbid physical or mental illness that is so impairing that they would be unable to participate in the groups or complete the measures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fear of cancer recurrence | Weeks 0, 6, 10, 30
  Multi-dimensional fear of recurrence measure.

SECONDARY OUTCOMES:
Anxiety | Weeks 0, 6, 10, 30
  Validated measure of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Laura B. Dunn, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States